CLINICAL TRIAL: NCT02996734
Title: Il Tumore a Cellule Giganti Delle estermità
Brief Title: Giant Cell Tumor of the Extremities Treated With Surgery and/or Medical Treatment
Acronym: GCTLIMBS
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Costantino Errani, MD; PhD., Istituto Ortopedico Rizzoli
Other Study IDs: 0008286
Record Dates: First submitted 2016-12-15; First posted 2016-12-19 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Giant Cell Tumor of Bone
Keywords: bone tumors; giant cell tumor; treatment
MeSH Terms: conditions — Giant Cell Tumor of Bone; Bone Neoplasms; Giant Cell Tumors | interventions — Curettage; Denosumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: curettage and resection — the investigators analyzed patients with giant cell tumor of bone who underwent curettage or resection with or without denosumab administration
  Other Names: denosumab

SUMMARY:
The purpose of this project is to present the outcomes of patients with giant cell tumor of bone (GCTB) who were treated with surgery and/or medical treatment in a single institution.

DETAILED DESCRIPTION:
The investigators retrospectively review patients treated for GCTB of the extremities between 1990 and 2013 in a single institution. We evaluate the recurrence free survival rate after surgical and medical treatment of patients with GCTB of the extremities to determine the influence of the surgical approach, denosumab therapy, local tumor presentation, and demographic factors on the risk of recurrence.

ELIGIBILITY:
Inclusion Criteria:

* giant cell tumors of the extremities

Exclusion Criteria:

* giant cell tumors of the spine and pelvis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with giant cell tumor of bone treated in a single institution
Sampling Method: Non-Probability Sample
Enrollment: 412 (Actual)
Dates: Start 2016-04; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
local recurrence rate after surgical and medical treatment | within the first 36 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Davide Donati, MD, Study Director — Istituto Ortopedico Rizzoli

IPD SHARING:
Plan to Share IPD: Yes
publish a manuscript in international medical journal

REFERENCES:
- [Derived] Tsukamoto S, Mavrogenis AF, Leone G, Righi A, Akahane M, Tanzi P, Kido A, Honoki K, Tanaka Y, Donati DM, Errani C. Denosumab does not decrease the risk of lung metastases from bone giant cell tumour. Int Orthop. 2019 Feb;43(2):483-489. doi: 10.1007/s00264-018-4085-6. Epub 2018 Aug 11. PMID 30099641